CLINICAL TRIAL: NCT03073928
Title: Comparison of Paracoracoid Subscapularis Plane Block to Interscalene Block for Arthroscopic Shoulder Surgery
Acronym: SPBvsISB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 108648
Record Dates: First submitted 2016-11-11; First posted 2017-03-08 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-06

CONDITIONS: Rotator Cuff Injury
Keywords: Nerve block; Diaphragm function
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Block (Active Comparator): Receives interscalene block with 15mL of ropivacaine 0.5% at the level of C6. A total of 15mL will be injected with repeated aspirations to rule out intravascular placement of the needle tip. Once this is done, the needle tip will be moved to the lateral edge of sternocleidomastoid muscle and additional 3mL of 0.5% ropivacaine will be injected between the deep fascia of the sternocleidomastoid and deep investing fascia of the neck (superficial cervical plexus block SCP).
  We will administer injection of saline similar to experimental group to blind the patient
  Interventions: Procedure: Interscalene Block; Drug: Ropivacaine
- Paracoracoid SPB (Experimental): Receives paracoracoid subscapularis plane block with the ultrasound. Using a 50mm 22G block needle 15ml of 0.5% Ropivacaine will be deposited anterior to the fascia of subscapularis muscle after eliciting a motor response with 0.6mA current delivered through the needle. Following this, superficial cervical plexus block will be done using 3mL of 0.5% ropivacaine similar to group 1.
  Interventions: Procedure: Paracoracoid SPB; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Interscalene Block — Regional Anesthesia procedure in the neck
  Arms: Interscalene Block
Procedure: Paracoracoid SPB — Regional anesthesia procedure under the collar bone
  Arms: Paracoracoid SPB
Drug: Ropivacaine — Amide local anesthetic Ropivacaine will be used in same concentration (milligrams) in both active comparator and experimental group

SUMMARY:
One hundred and twenty patients will be randomized to Interscalene block or Paracoracoid Subscapularis plane block. The study will evaluate the efficacy and duration of blocks in the 2 groups with regards to postoperative analgesia and degree of respiratory depression.

DETAILED DESCRIPTION:
Background:

Postoperative pain after arthroscopic shoulder surgery can be severe in 30- 70% of the patients in the first twenty-four to forty-eight post-operative hours . Single injection interscalene block (ISB) is commonly offered to decrease postoperative pain following shoulder surgery with many associated benefits like reduced opioid consumption, nausea and decreased Postoperative Acute Care Unit (PACU) stay. The adverse events of the ISB may be reduced with ultrasound guidance but are not completely eliminated. One of the major concerns is the phrenic nerve involvement resulting in diaphragm paresis, which has major implication in patients with respiratory compromise. One of the alternatives is blockade of the suprascapular nerve in the suprascapular fossa and the axillary nerve as it curves around the humeral neck. Although researchers from Australia have reported a good outcome with it an earlier study done by us had a suboptimal effect (102994), possibly because the nerves were blocked after the articular branches had exited the main trunk.

There are studies currently ongoing with blocks being done more proximally in our center but that requires 2 injections. The investigators did an anatomical study on Fresh frozen cadavers and noted that drugs delivered superficial to the Fascia of Subscapularis muscles stains the Axillary Nerve, Upper subscapular nerve and possibly suprascapular nerve before it enters the suprascapular fossa

The extent to which the two techniques differ in terms of overall analgesia has not been evaluated. With this background, The investigators want to compare the analgesic efficacy of interscalene block versus Paracoracoid Subscapularis plane block when combined with superficial cervical plexus block.

Aims and objectives:

The objective of the study is to compare the efficacy and safety of the paracoracoid subscapularis plane block with interscalene block to control pain after arthroscopic shoulder surgery. The primary outcome will be duration of analgesia provided by the regional blocks. The duration is defined as the time from the end of injection of local anesthetic to the time when patient requests rescue analgesia (pain score greater than 6 out of 10). The secondary outcomes include measurement of degree of respiratory depression via Pulmonary Function Test and ultrasound assessment of diaphragmatic function, first 24 and 48th hour pain scores, time needed to perform each type of block, and post-operative opioid requirement (24 hour analgesic consumption) and the failure rate.

Primary Hypothesis:

Paracoracoid Subscapularis plane block results in comparable analgesia to interscalene blocks sparing the Phrenic nerve

Secondary hypothesis:

1. Paracoracoid Subscapularis Plane block results in better preserved diaphragm function compared to interscalene block.
2. The failure rate is similar between the two groups (null hypothesis)
3. The postoperative opioid consumption is similar between the 2 groups (null hypothesis)

Methodology:

After institutional approval and informed consent, 120, patients of either sex belonging to American Society of Anesthetists (ASA) physical status 1 to 3 scheduled for elective arthroscopic shoulder surgery will be included in the study. Patients receiving chronic narcotic therapy, patients with major respiratory morbidity, morbid obesity or patients with peripheral neuropathies and who cannot provide an informed consent will be excluded from the study. Patients will be educated regarding the numerical rating score (NRS) on a scale of 0 to 10 where 0 is no pain and 10 is the worst pain ever experienced and their preoperative NRS scores will be documented.

Patients will be randomized into one of 2 groups using a web based randomization. All procedures will be done in the block room using sterile precautions, standard monitors and intravenous sedation as per the standard practice at our hospital. The baseline respiratory function will be measured with bedside spirometry, which will be repeated at 3 time points: Pre block, 20 minutes post block and about 60 minutes after arrival in the PACU post-surgery. Patients diaphragm thickness will be measured on both sides of the chest, with the patient seated, at the anterior axillary line using a high frequency linear probe positioned vertically and the position of the probe will be marked on the skin on both sides to ensure comparable measurements. Patients will be asked to take a big breath 3 times+/-sniffs and loops of diaphragm movements will be recorded on the ultrasound machine. The point where the diaphragm peels off from the chest wall will be noted on the ultrasound and the thickness of the diaphragm will be measured using the caliper available on the US machine. The thickness will be averaged out between 3 measurements. These measurements will be repeated on the contralateral side. Once this is completed, patients will be connected to the standard monitors (EKG, Pulse oximetry and NIBP) and they will receive supplemental oxygen. All patients will receive titrated doses of intravenous fentanyl and midazolam for conscious sedation as per the standard practice at our institution. All patients will be positioned supine with 45 degree head up tilt with a rolled blanket under the ipsilateral side to allow slight rotation to the contralateral side.

Group 1 will receive interscalene block with 15mL of ropivacaine 0.5% at the level of C6 ventral ramus as identified with the 7-12MHz linear probe positioned horizontally. Neurostimulation with 0.6mA should result in contractions of the deltoid and biceps. A total of 15mL will be injected with repeated aspirations to rule out intravascular placement of the needle tip. Once this is done, the needle tip will be moved to the lateral edge of sternocleidomastoid muscle and additional 3mL of 0.5% ropivacaine will be injected between the deep fascia of the sternocleidomastoid and deep investing fascia of the neck (superficial cervical plexus block SCP). The start and finish time will be recorded. In addition, probe will be moved similar to the group two and skin infiltration with saline will be done to blind the patient.

Group 2 will receive paracoracoid subscapularis plane block with the ultrasound probe positioned on the head of the humerus in the sagittal plane. The probe is then moved medial to locate the coracoid process. Pectoralis major, pectoralis minor and subscapularis muscle in the scapular fossa are identified. Using a 50mm 22G block needle 15ml of 0.5% Ropivacaine will be deposited anterior to the fascia of subscapularis muscle after eliciting a motor response with 0.6mA current delivered through the needle. Following this, superficial cervical plexus block will be done using 3mL of 0.5% ropivacaine similar to group 1. All patients will receive a small band-aid in the 2 locations of possible needle entry to blind the observer to the randomization.

An independent observer will document the motor and sensory block 20 minutes after the block injection is completed for each group. Patients will then have a bedside spirometry repeated. They will be in the sitting position. Ultrasound evaluation of the diaphragm will be done bilaterally at the anterior axillary line posteriorly positioning the probe exactly where it had been marked pre-block. The thickness of the diaphragm will be assessed using an average from three deep inspirations/sniffs.

Total duration of block performance, number of attempts for block and the time for the onset of sensory block will be recorded after the performance of the block, by a blinded observer. The failure rate of nerve block will be determined by the blinded observer at 30 minutes. Patients with failed blocks will be excluded from the efficacy part of the study. After performance of the blocks, the patient will be moved to the operating room for the surgery under general anesthesia according to the choice of the anesthesiologist (LMA vs. endotracheal intubation) using fentanyl 2-3µg/Kg, propofol 2 mg/kg followed by maintenance with desflurane/sevoflurane in air-oxygen mixture. Vasopressors and opioids will be administered as needed titrated to the clinical effect. Total dose of narcotic used will be recorded. The patients will be assessed for the site and severity of pain at rest and movement after arrival in the PACU and at 2 hourly intervals till discharge from PACU. Patients will be provided with a diary to document pain scores every 6 hourly thereafter until 24 hours after their time of arrival in PACU (time 0). Patients will be contacted by one of the investigators to ensure that their pain is well controlled and to get their pain scores and ongoing narcotic consumption at 9PM day of surgery and at 7AM on postoperative day 1. They will be reminded to fill in the data sheet and to mail it back to us. The investigators will inquire about the precise time point of when the block wore off. The investigators will also seek information about persisting neurological deficits at the 7AM call. If pain is severe (>7/10) on arrival to PACU, it will be defined as failure of the technique and they will be given intravenous hydromorphone 0.2-0.4mg titrated to effect in the PACU. An emergency telephone number will be provided in case of any medical problems until 24 h after performance of the blocks. All patients will be followed up 24 and 48 hours later to find out if there are any persisting neurological deficits as per the standard practice at our institution. The investigator at this point will collect data regarding duration of block, time to first rescue analgesia, total analgesic requirement and occurrence of any complications related to nerve block. Patients will be given instructions during this call to contact us if they develop new onset neurological deficits/symptoms in the following 4 weeks. Patient satisfaction will be documented at 24 hours on a visual analogue scale where 0 is totally dissatisfied and 100 is totally satisfied. The total participation time for the patients is for 2 days.

Statistical Analysis:

Data will be presented as the mean +/- SD and median (min, max) for all continuous data including duration in hours, respiratory function, pain, and patient satisfaction at all time points for both groups. Statistical comparisons between-group will be made using an ANCOVA where block group is the fixed effect, the endpoint is the dependent variable and the pre-block score is the covariate. This will produce an adjusted mean between-group difference with 95%CI. The adjustment by pre-block score will also providing a more precise estimate of the effect. If the lower boundary of the 95%CI from the adjusted mean difference for duration is greater than 2 hours the investigator will declare that the SPB is superior to the ISB. Because it will be of interest to institutions in terms of resource use and cost, the procedure-related data like time to administer each block, time to sensory onset, total narcotic dose, and number of attempts will be presented using mean +/-SD, median (min, max) and mean difference with 95%CI. Nominal data like failure rate and complications will be described using proportions. Site and severity of pain at rest and with movement will be presented using line graphs to support hypothetical expected locations of pain given what the investigator know about anatomical innervation related to the type of block administered.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 16-85years of age, scheduled to undergo arthroscopic shoulder surgery.
2. Elective shoulder surgery undergoing general anesthesia in combination with regional blockade.
3. ASA Class I,II and III
4. Able to give informed consent
5. Able to cooperate with study process
6. Availability of home telephone

Exclusion Criteria:

1. ASA 4
2. Refusal to have regional block
3. Lack of informed consent.
4. Language or reading barrier
5. Allergy to any of the drugs used in the study.
6. Patients with associated significant cardiac and respiratory disease.
7. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
8. Patients with coexisting hematological disorder or with deranged coagulation parameters.
9. Significant psychiatric illnesses. (Schizophrenia or bipolar disorders, uncontrolled anxiety or depression)
10. Narcotic dependency (Chronic opioid use of greater than 15 mg oral morphine equivalents daily)
11. Peripheral neuropathy
12. Pregnancy
13. Emergency surgery

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | Pain NRS measured every 120 minutes until score of 6/10 is obtained (up to 24 hours).
  Duration in hours from end of injection to patient reported pain NRS score of more than 6/10

SECONDARY OUTCOMES:
Measurement of diaphragm thickening pre and post block | 3 measurements - pre block, 20 minutes post block & 1 hour post surgery
  Measurement of diaphragm thickening pre and post block using ultrasound

OTHER OUTCOMES:
Measurement of Forced Expiratory Volume in 1 second (FEV1) | 3 measurements - pre block, 20 minutes post block & 1 hour post surgery
  Measurement of FEV1 to assess pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Sugantha Ganapathy, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, St. Joseph's Heath Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sondekoppam RV, Lopera-Velasquez LM, Naik L, Ganapathy S. Subscapularis and sub-omohyoid plane blocks: an alternative to peripheral nerve blocks for shoulder analgesia. Br J Anaesth. 2016 Dec;117(6):831-832. doi: 10.1093/bja/aew370. No abstract available. PMID 27956687